CLINICAL TRIAL: NCT05634330
Title: The Effect of Core Stabilization Exercises on Balance and Quality of Life in Chronic Period in Individuals With Lumbar Disc Herniation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Asiye Uzun, Principal investigator, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HasanKU AU-001
Record Dates: First submitted 2022-10-15; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Lumbar Disc Herniation; Balance; Distorted
Keywords: Lumbar Disc Herniation,; Chronic Period, Balance,; Core Stabilization,; Proprioceptive Sense
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Intervention Model Description: two group. one of group for exercise and the other group is for control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): treatment group: core stabilization exercises used to improve balance
  Interventions: Other: exercise treatment
- control group (No Intervention): this group members have continued their normal lives

INTERVENTIONS:
Other: exercise treatment — core stabilization exercise
  Arms: treatment group

SUMMARY:
The Effect of Core Stabilization Exercises on Balance and Quality of Life in Chronic Period in Individuals With Lumbar Disc Herniation

DETAILED DESCRIPTION:
This study was carried out to examine the effect of core stabilization exercises on balance and quality of life in the chronic period in individuals with lumbar disc herniation. Forty patients aged 45-65 years who had been diagnosed with lumbar disc herniation at least one year ago were included in the study. By randomization, they were divided into 2 groups of 20 people, each being the treatment and the control group. A self-prepared form for patient demographic information, McGill Pain Scale and Visual Analog Scale(VAS) for pain assessment; Diasu Gait Analysis Device and Berg Balance Scale for static balance assessment; Timed Up and Go Test, Y Balance Diagram, Functional Reach Test to evaluate dynamic balance; Tinetti Fall Efficiency Scale for assessing falls; The Oswestry Disorder Scale and Nottingham Health Profile were used to assess quality of life and functionality; to evaluate proprioceptive sensation, ankle joint position sense was measured in standing, neutral position (0˚) and angular measurement in 10˚ dorsiflexion. After the questionnaires and measurement tools were completed, the patients were included in the program. While the patients in the control group continued their routine lives, the modified pilates exercise program focused on core stabilization was applied to the patients in the treatment group for 8 weeks, 2 days a week for 50 minutes and in 4 groups. After the treatment process was completed, the questionnaires and measurements were repeated.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 45 and over with a diagnosis of Lumbar Disc Herniation,

  * Not having any communication barriers (sight, hearing, hearing),
  * Have not undergone any surgical procedure in the last 6 months,
  * Patients who volunteered to participate in the study

Exclusion Criteria:

* Those who do not want to participate in the study,

  * Individuals whose age is unsuitable,
  * Individuals who continue to receive a therapeutic exercise therapy,
  * Individuals with a neurological condition that may affect ankle muscle strength and sensation

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in static balance on Diasu Gait Analysis Device at Week 8 | baseline and Week 8
  To evaluate static balance looking at oscillation length in 1 minute Change= (Week 8 score - Baseline score)
Change from baseline in weight bearing on Diasu Gait Analysis Device at Week 8 | baseline and Week 8
  To evaluate weight bearing looking at weight percent for each foot Change= (Week 8 score - Baseline score)
Change from baseline in static and dynamic balance on Berg Balance Test at Week 8 | Baseline and Week 8
  To evaluate static and dynamic balance. It consists of evaluating 14 activities implemented by direct observation of performance. Each item is scored between 0-4. 0 represents the worst and 4 the best. The total highest score is 56. Scores of 45 and below indicate a risk of falling.
  Change= (Week 8 score - Baseline score)
Change from baseline in dynamic balance and functionality on Timed Up and Go Test at Week 8 | Baseline and Week 8
  To evaluate dynamic balance and functionality. The person is asked to get up from the stool, to walk with a safe and normal walking speed, to turn and to sit on the stool again. The distance between two stools is fixed at 3 meters. The application time is recorded in seconds. A shorter duration indicates better balance and mobility.
  Change= (Week 8 score - Baseline score)
Change from baseline in dynamic balance and functionality on Y Balance Test at Week 8 | Baseline and Week 8
  To evaluate dynamic balance and functionality. While standing on one foot, he is asked to take steps with the other foot first anteriorly, then posterolaterally, and finally in the posteromedial direction. At this time, care must be taken that the foot on the ground does not rise from the ground and the balance is not disturbed. The test is repeated 3 times in each direction and the average is taken and recorded in cm. The same measurement is applied to the other foot in the same way.
  Change= (Week 8 score - Baseline score)
Change from baseline in dynamic balance and functionality on Functional Reach Test at Week 8 | Baseline and Week 8
  To evaluate dynamic balance and functionality. The individual is asked to stand upright for the test and to extend the arm to be measured forward. As the starting point, the 3rd fingertip strip is brought to the 0 point on the tape measure. The tape measure is fixed by the physiotherapist and the patient is asked to lie on the tape measure without losing the contact of the feet with the ground. The test is repeated 3 times and the best distance is recorded in cm. The test is repeated 3 times and the best distance is recorded in cm for the right and left measurement.
  Change= (Week 8 score - Baseline score)
Change from baseline in dynamic balance and for assessing falls on Tinetti Fall Efficiency Scale at Week 8 | Baseline and Week 8
  To evaluate dynamic balance and for assessing falls. It is a questionnaire consisting of 10 questions measuring A score between 1-10 is given. 1 is scored as very safe and 10 is scored as very high fear of falling. The total highest score is recorded as 100.
  Change= (Week 8 score - Baseline score)
Change from baseline in pain on Mcgill pain Scale at Week 8 | Baseline and Week 8
  To evaluate pain degree. It is a questionnaire that questions the severity of the pain, its location, its first relationship over time, the sensation it creates in people, and whether it is livable pain for individuals.
  Change= (Week 8 score - Baseline score)
Change from baseline in pain on Visual Analog Scale at Week 8 | Baseline and Week 8
  To evaluate pain degree. A score between 0-10 is given. 0 means no pain and 10 is scored as excruciating pain.
  Change= (Week 8 score - Baseline score)
Change from baseline in proprioceptive sensation on ankle joint position sense at Week 8 | Baseline and Week 8
  To evaluate proprioceptive sensation, ankle joint position sense was measured in standing, neutral position (0˚) and angular measurement in 10˚ dorsiflexion.
  Change= (Week 8 score - Baseline score)
Change from baseline in quality of life and functionality on Nottingham Health Profile at Week 8 | Baseline and Week 8
  To assess quality of life and functionality. It is a scale that questions psychological well-being from different aspects such as physical activity, pain, emotional state, sleep, social life, energy. Short answers are given as yes or no. A person can get a maximum of 600 points. An increase in the score obtained means that the level of quality of life decreases.
  Change= (Week 8 score - Baseline score)
Change from baseline in quality of life and functionality on Oswestry Disorder Scale at Week 8 | Baseline and Week 8
  To assess quality of life and functionality. It is a questionnaire consisting of 10 items. The person can get points between 0-10 from each item. 0 represents the best level and 5 represents the worst level. The total score is a maximum of 100. As the score increases, it is shown that the functionality of the person worsens and the level of disability increases.
  Change= (Week 8 score - Baseline score)
A self-prepared form | Baseline
  For patient demographic information,

CONTACTS AND LOCATIONS:
Locations (1):
- As Physiotherapy Office, Gaziantep, Gazi̇antep, Turkey (Türkiye)